CLINICAL TRIAL: NCT01182987
Title: SCAN Memory Program Evaluation Study
Acronym: SMPES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Joshua Chodosh, MD, MSHS / Principal Investigator, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: SRC 09-002
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Dementia
Keywords: Quality improvement; Quality of care; Health care utilization; Behavioral change
MeSH Terms: conditions — Dementia; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dementia care management (Active Comparator): Patients and family caregivers will be offered dementia care management, which includes detailed comprehensive assessment, education, counseling, referrals to community agencies, collaboration with medical providers and frequent telephone follow-up
  Interventions: Behavioral: Dementia Care Management
- Usual care (No Intervention): Patients and care family care givers will receive usual support and medical care offered by the health plan.

INTERVENTIONS:
Behavioral: Dementia Care Management — The SCAN Memory Program is a care management program for cognitively-impaired SCAN members and for their informal/family caregivers. The program includes collaboration between SCAN Health Plan, partnering medical groups, and community organizations.
  Program activities include: 1) telephonic-structured assessments with informal caregivers conducted by SCAN Memory Program care managers; 2) problem identification as a result of these assessments; and 3) pre-established protocols and procedures for problem resolution.
  Arms: Dementia care management

SUMMARY:
The SCAN Memory Program Evaluation study is an evaluation of a randomized controlled trial intervention consisting of a care management program for cognitively-impaired health plan members and for their informal/family caregivers. The program includes collaboration between the health plan, partnering medical groups, and community organizations.

Program activities include: 1) telephonic-structured assessments with informal caregivers conducted by SCAN Memory Program care managers; 2) problem identification as a result of these assessments; and 3) pre-established protocols and procedures for problem resolution. ACCESS, the prototype for the SCAN Memory Program, was developed and tested in San Diego County and was very successful in helping affected patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria: Health plan member eligibility includes having a visit-based ICD-9 diagnostic code for dementia or a dementia-specific medication (including donepezil, rivastigmine, galantamine, and memantine) within administrative data any time prior to data inquiry for potential subjects. The health plan member must have a caregiver who can communicate by telephone and though that person might also be a health plan member, health plan membership for caregivers is not required. All subjects must be living in the community and if in a nursing facility, this must be for rehabilitation or respite care but not for long term care. Caregivers must be able to communicate in English or Spanish.

Exclusion Criteria: Person with dementia whose potential participation is declined by their physician. Those who do not have a family or informal caregiver cannot participate and caregivers who do no have telephone access or the capacity to consent to research evaluation are excluded. Patients who reside in nursing facilities as permanent residents are not eligible.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Guideline Adherence | 18 months of longer
  Quality of care process measures will be examined that reflect practice guideline quality indicators measuring patient and caregiver assessment, treatment, education and support, and safety. Measures are collected at 9 and 18 months using caregiver surveys and medical record abstraction.
Program feasibility and fidelity | 6 to 18 months
  Formative Evaluation consisting of a series of stakeholder semi-structured interviews and data abstraction to monitor the activities of healthplan care managers will be collected at pre-specificed intervals and results will be provivided periodically to the healthplan for ongoing improvements in program delivery.
Healthcare utilization | 18 months
  Caregiver specific utilization including use of services that care managers may recommend to them and the dementia patient. Emergency department, hospitalization and ambulatory visits data will also be collected through administrative data and caregiver surveys.

SECONDARY OUTCOMES:
Behavioral disturbance | 9 months and 18 months
  Neuropsychiatric inventory questionnaire (NPI-Q)as a caregiver derived assessment on caregiver surveys conducted at baseline, 9 and 18 months.
Functional Status | 9 and 18 months
  Using an informant (caregiver)-based measure of 10 complex higher order activities using the Functional Activities Questionnaire (FAQ). This is a reliable measure of functional status in patients with dementia.
Quality of life | 9 and 18 months
  Patient health related quality of life (HRQOL) using the Health Utilities Index
Quality of Care | 9 and 18 months
  Using caregiver surveys, this will be measured with a 5-item scale from the Consumer Assessment of Health Plans Survey 2.0.
Caregiver self-efficacy | 9 months and 18 months
  caregiver confidence using a 6-item measure that was utilized in prior care management clinical trials
Caregiver unmet need for assistance | 9 months and 18 months
  a 2-item, 3-point scale for each covering general caregiveing - bathing, dressing, and transportation
Caregiver social support | 9 months and 18 months
  This will be measured in caregiver surveys using a 5-item measure derived from the Medical Outcomes study Social Support Survey (MSSS).
Caregiver burden | 9 months and 18 months
  The 22-item Burden Interview is a widely used validated measure to assess stressors experienced by caregivers of persons with dementia. Each itme uses a 5-point scale (response set).
Caregiver depression | 9 months and 18 months
  The Patient Health Questionnaire - Nine (PHQ-9) will be included in caregiver surveys at baseline, 9 and 18 months as a measure of depressive symptoms over the preceding 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD, MSHS, Principal Investigator — VA / UCLA
Locations (2):
- United States (2):
  - Davis Research, Calabasas, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California